CLINICAL TRIAL: NCT01419756
Title: Assessment of Right Ventricular Volume Using the Ventripoint Medical System in Patients With Tetralogy of Fallott Following Repair; A Comparison Study to cMRI
Brief Title: Assessment of Right Ventricular Volume in Tetralogy of Fallott (TOF) Patients
Acronym: VMS TOF
Status: Completed | Type: Observational
Sponsor: VentriPoint Diagnostics Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2011041
Record Dates: First submitted 2011-08-16; First posted 2011-08-18 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2013-07

CONDITIONS: Tetralogy of Fallot
MeSH Terms: conditions — Tetralogy of Fallot

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single Arm: Imaging comparison study. No intervention.
  Interventions: Device: VentriPoint Medical System

INTERVENTIONS:
Device: VentriPoint Medical System — The Knowledge Based Reconstruction (KBR) method generates a 3D reconstruction of the RV based on the Piecwise smooth subdivision surface method but without requiring manual border tracing. Instead KBR reconstructs a new patient's ventricular surface from the placement of anatomic landmark points on a 2D ultrasound image

SUMMARY:
Assessment of Right Ventricular Volume using the VentriPoint Medical system in patients with Tetralogy of Fallot following repair; a comparison study to cMRI.

The objective of this study is: To evaluate the accuracy of the VentriPoint Medical System to calculate right ventricular volumes in patients with Tetralogy of Fallot following surgical repair.

Secondary objectives are: To validate Inter and Intra observer variability at 3 clinical sites.

The analyses will be the same for EDV and ESV. For either right ventricular volume, the primary effectiveness measure is the % difference between VMS and cMRI results, i.e. (VMS-cMRI)*100%/average of VMS and cMRI results. There will be two null hypotheses for the primary analysis:

H0+: true mean % difference > 10% and H0-: true mean % difference < -10%

The observed mean % difference will be presented with 95% confidence intervals. The VMS right ventricular volume estimates will be regarded as equivalent to cMRI estimates if both H0+ and H0- are rejected at a 1-sided 0.025 level by a paired t test for both EDV and ESV. Since H0+ and H0- cannot both be true, the total type I error rate for each measure is 0.025 and the overall type I error rate for both EDV and ESV is 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Tetralogy of Fallot following surgical repair
* Patients who can be expected to lie motionless during imaging

Exclusion Criteria:

* Lack of informed consent
* Surgical repair for Tetralogy of Fallot with RV-PA conduit
* Known arrhythmia that interferes with image acquisition.
* Implanted cardiac defibrillator, pacemaker, or other devices containing ferromagnetic materials
* Pregnant woman
* Contraindications for MRI

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary Care Clinic Cardiac Clinic
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2011-08; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of this study is the percent difference between the VentriPoint Medical System (VMS) and cMRI for estimating the end diastolic and end systolic right ventricular volumes (EDV and ESV) in subjects following repair for TOF. | 4 months
  The trial will be regarded as successful if it demonstrates the mean VMS-cMRI percent difference to be <10% and >-10% at a 1-sided 0.025 statistical significance level for each of EDV and ESV, with no safety concerns for the VMS procedure.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (5):
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Cleveland Clinic, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Children's Hosptial of Philadelphia, Philadelphia, Pennsylvania
- Hospital for Sick Children, Toronto, Ontario, Canada